CLINICAL TRIAL: NCT05436548
Title: The Work-life Check-ins: a Supervisor-driven Intervention to Reduce Burnout in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Hurtado, ScD, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020965
Record Dates: First submitted 2022-06-21; First posted 2022-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Burnout
Keywords: burnout; values alignment; supervisor support
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Primary care clinics randomly assigned to the intervention will conduct frequent supervisor-employee check-ins. Supervisors at those clinics will receive training to conduct such check-ins. Control clinics will continue as usual practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief and frequent Work-life check-ins between clinic supervisors and each staff member (Experimental): Primary care clinics assigned to the intervention will conduct frequent (every 8 weeks) supervisor-employee brief (30 min) check-ins to identify work stressors. Supervisors at such clinics will complete training on how to use the check-ins to address work stressors.
  Interventions: Other: Supervisor-employee frequent check-ins to identify and address work stressors
- Usual practice, waitlist controls (Experimental): Primary care clinics randomly assigned to the control condition will continue as usual practice. If the check-is are effective in reducing burnout, then supervisor-level training will become available to supervisors at the end of the study
  Interventions: Other: Usual practice waitlist controls

INTERVENTIONS:
Other: Supervisor-employee frequent check-ins to identify and address work stressors — Supervisors will complete three training modules: 1) how and why the check-ins are expected to address burnout; 2) how to demonstrate supportive supervision during the check-ins process, and 3) principle of quality improvement applied to the check-ins
  Arms: Brief and frequent Work-life check-ins between clinic supervisors and each staff member
Other: Usual practice waitlist controls — If the check-ins are successful in reducing burnout, supervisors at the control clinics will be offered the training modules
  Arms: Usual practice, waitlist controls

SUMMARY:
The objective of this study is to evaluate the effectiveness and process of frequent supervisor-employee check-ins in reducing burnout among employees of primary care clinics in Portland, OR. Healthcare workers are at risk for burnout and associated adverse health and safety outcomes, including chronic diseases and occupational injuries. Not only does burnout affect healthcare workers, but burnout also affects the quality of patient care. The proposed study will create a check-in process between supervisors and healthcare workers, which addresses supervisor support, awareness of services and resources, and work-life balance. The Work-life Check-ins project expects to see reduced burnout among employees participating in the check-ins intervention compared to those in the control group.

DETAILED DESCRIPTION:
Burnout is a manifestation of chronic work stress characterized by emotional exhaustion, cynicism, and diminished self-efficacy. The burden of burnout is alarming, especially within healthcare where it affects at least one-third of the workforce, including clinicians and support staff. The causes of healthcare worker burnout are multifactorial, including systemic pressures (e.g., intensification of charting duties, prolonged work hours with circadian and work-life disruptions, exposure to trauma), and unit-level characteristics (e.g., value misalignment and mistrust between team members and leadership, and lack of supportive services or resources). The modification of these systemic factors requires the lengthy action of stakeholders that have competing agendas. In the meantime, the healthcare workforce remains in urgent need of practical, adaptable, and meaningful solutions to start addressing this pervasive problem. In this conundrum, interventions aimed at improving leader-staff relations - a more readily modifiable target than systemic pressures- have reduced the most proximal emotional effects of burnout. However, new approaches are required so that leadership-focused interventions generate and sustain impactful organizational transformations. The need for such interventions is even more significant amid the exploding levels of work stress related to the COVID-19 crisis.

The objective of this five-year proposal is to conduct a cluster randomized controlled trial (CRT) across 10 OHSU primary care clinics to evaluate the effectiveness and process of a supervisor-focused intervention to reduce burnout. The intervention titled "Work-life Check-ins" will create a process designed to reduce burnout by boosting supervisor support, trust, and value alignment, increasing awareness of appropriate services and resources, and addressing workflow or work-life problems. The central hypothesis is that employees at the six clinics randomly assigned to the intervention will have reduced burnout at the 12- month follow-up compared to waitlist-control clinics. The investigators expect that the intervention will reduce burnout based on our preliminary studies and the integration of evidence-based techniques, including supportive supervision training, goal setting, feedback sessions, and quality improvement cycles. This proposal will accomplish the following specific aims.

Aim 1: Determine the Work-life Check-ins' effectiveness on burnout and secondary outcomes.

The investigators will evaluate the effectiveness of the Work-life Check-ins via surveys conducted among eligible employees (N=552 across the 10 clinics). As the primary outcome, it will be surveyed burnout at baseline and after 12 months. As secondary outcomes, we will examine safety and well-being variables (e.g., turnover intentions, values alignment, supervisor support and safety climate,).

Aim 2: Identify organizational changes produced by the Work-life check-ins. The investigators will conduct a multi-method process evaluation, including implementation metrics (e.g., number and frequency of check-ins) and in-depth interviews with supervisors and workers after implementation. The process evaluation will reveal the extent to which the intervention influenced the adoption of environmental, procedural or educational burnout control and prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Employed at one of the 12 OHSU primary care clinics that weren't involved in the pilot study
* Supervisors (medical director, practice manager, supervisors, leads)
* Employees (patient-facing; back and front of the clinic)

  * Patient Access Specialists
  * Medical Assistants
  * MDs, RNs, NPs

Exclusion Criteria:

* Under the age of 18
* Employed at an OHSU primary care clinic that participated in the pilot study
* Non-clinic employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Burnout baseline vs. 12th month follow-up | 12 months post supervisor check-ins training
  As a primary outcome, we will use the Maslach Burnout Inventory, which is considered the gold standard in burnout research. The MBI-HSS yields a three-factor score of burnout: emotional exhaustion (9 items; e.g., "I feel burned out from my job"), depersonalization (5 items; e.g., "I've become more callous toward people since I took this job"), and low personal accomplishment (8 items; "I feel I'm positively influencing other people's lives through my job).

SECONDARY OUTCOMES:
Change in Turnover intentions baseline vs. 12th month follow-up | 12 months post supervisor check-ins training
  We will measure turnover intentions as the average of two questions, scored with a 5-point scale (NIOSH Quality of Work Life), about the extent to which participants are considering leaving their current job and organization (higher scores means higher intentions).
Change in Values alignment with clinic leaders baseline vs. 12th month follow-up | 12 months post supervisor check-ins training
  The Mini-Z has 10 questions (continuous variables) for aspects such as value alignment (e.g., "my professional values are well aligned with those of my clinic leader"). Higher scores means higher values alignment.
Change in Family Supportive Supervisor Behaviors (FSSB) baseline vs. 12th month follow-up | 12 months post supervisor check-ins training
  The study will include a modified version of the Family-supportive supervisor behaviors (FSSB) questionnaire, created by Dr. Hammer. The FSSB has 4 questions for emotional support, instrumental support, role modeling and creative conflict management (e.g., "my supervisor works effectively with employees to solve conflicts between work and non-work creatively"). Higher scores means higher FSSB.
Change in Organizational constraints baseline vs. 12th month follow-up | 12 months post supervisor check-ins training
  Organizational constraints is a scale that inquires the extent to which workers perceive that different barriers affect their performance. This scale (title: Organizational Constraints Scale) asks about equipment, supplies, procedures, supervisors, co-workers, insufficient training, and incorrect instructions, among others (11 items; e.g., "how often do you find it difficult or impossible to do your job because of"). Higher scores mean greater constraints.

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurtado DA, Boyd J, Madjlesi R, Greenspan SA, Ezekiel-Herrera D, Potgieter G, Hammer LB, Everson T, Lenhart A. The Work-life Check-ins randomized controlled trial: A leader-based adaptive, semi-structured burnout intervention in primary care clinics. Contemp Clin Trials. 2024 Aug;143:107609. doi: 10.1016/j.cct.2024.107609. Epub 2024 Jun 13. PMID 38878996